CLINICAL TRIAL: NCT00113347
Title: Phase I Evaluation of Erlotinib and Docetaxel With Concomitant Boost Radiation for Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Erlotinib and Docetaxel With Concomitant Boost Radiation Therapy (XRT) for Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-1049
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Squamous Cell Carcinoma; Erlotinib; Docetaxel; Radiation; Radiotherapy; Concomitant Boost Radiation
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Erlotinib Hydrochloride; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib + Docetaxel (Experimental): Erlotinib 100, 125, or 150 mg orally daily except days receive Docetaxel 15 mg/m^2 or 20 mg/m^2 intravenously with Concomitant Boost Radiation to Head/Neck
  Interventions: Drug: Erlotinib; Drug: Docetaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Erlotinib — Beginning on Day 2 of treatment, 100, 125, or 150 mg by mouth once a day every day while on treatment, except on days docetaxel is received.
  Other Names: Tarceva; OSI-774; Erlotinib Hydrochloride
Drug: Docetaxel — 15 mg/m^2 or 20 mg/m^2 by vein over 15 to 30 minutes on Days 1, 8, 15, and 22 of treatment.
  Other Names: Taxotere
Radiation: Radiation Therapy — Radiation therapy to head/neck beginning on day 1 of treatment once daily 5 times per week (Monday through Friday), delivered in 40 fractions.
  Other Names: XRT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of the drugs OSI-774 and docetaxel that can be given together along with radiation treatment for advanced head and neck cancer.

DETAILED DESCRIPTION:
OSI-774 (also known as Erlotinib or Tarceva) is a drug that helps to block the activity of an enzyme that is believed to play an important role in cell growth. It is hoped that blocking this enzyme will slow tumor growth. Docetaxel (Taxotere) is a commonly used chemotherapy drug. Docetaxel is designed to target and destroy cancer cells.

Before beginning treatment, you will have a complete physical exam. You will also have routine blood (about 4 teaspoons) and urine tests, a chest x-ray or CT scan, and an electrocardiogram (ECG - test to measure the electrical activity of the heart). You will have a dental exam performed by a dentist. Women who are able to have children must have a negative pregnancy test (blood or urine). You will also have either a CT scan or a MRI to measure your disease. You may have a bone scan and/or CT scans of your abdomen and chest if your doctor thinks it is necessary for your care.

You will have a swallowing evaluation. The swallowing evaluation involves drinking barium and other liquids of varying thickness while fluoroscopy (like an x-ray movie) is done to evaluate swallowing function. You will also complete a questionnaire that asks questions about quality of life issues. The questionnaire should take about 10 minutes to complete.

In this study you will receive radiation therapy 5 days per week (Monday through Friday) for 6 weeks. You will not receive radiation therapy on weekends. For the first 3 weeks of treatment you will receive radiation once a day. Starting on the 4th week of treatment, you will receive radiation treatment twice a day. The treatments will be at least 6 hours apart. You will receive these twice daily radiation treatments Monday through Friday for 3 weeks.

On your first day of radiation treatment you will also receive your first dose of docetaxel. You will receive docetaxel by vein over 15 to 30 minutes on Days 1, 8, 15, and 22 of treatment.

Beginning on Day 2 of treatment, you will begin taking OSI-774 by mouth. You will take OSI-774 once a day in the morning with up to 7 ounces of water either 2 hours after or 1 hour before eating. If you are unable to swallow the OSI-774, you may dissolve it in distilled water and take it through a feeding tube. You will take OSI-774 every day while on treatment except on days on which you receive docetaxel (i.e., Days 1, 8, 15, and 22). You should not take OSI-774 on days you receive a docetaxel infusion.

Participants will enter this study in groups of 3. The doses of both OSI-774 and docetaxel will be increased after each group. Six patients will be studied at the dose level that is estimated to be the highest safe dose.

While receiving treatment on this study, you will be examined at least once a week. You will also have weekly blood tests (2-4 teaspoons). At the end of treatment, you will have another CT scan or MRI to measure your disease. You will also have a complete physical exam and blood tests (4 teaspoons). You may be taken off study if your disease gets worse or intolerable side effects occur.

After completing treatment, you will have a follow-up visit every 3 months for 2 years, then every 4 months during Year 3, and every 6 months during Years 4 and 5. These visits will include a medical history and physical exam. A CT or MRI study and blood work (2-4 teaspoons) may also be done. You will have swallowing evaluations at 3 and 12 months following treatment, and then once yearly through year 5. When you have these swallowing evaluations, you will also be asked to complete a short questionnaire about swallowing. The questionnaire will take about 10 minutes to complete.

This is an investigational study. OSI-774 is approved by the FDA for treatment of non-small cell lung cancer. Docetaxel is approved by the FDA for treatment of lung cancer and breast cancer. Their use together in this study with radiation treatment is experimental. Up to 24 patients are expected to take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological proof (from the primary lesion and/or lymph nodes) of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx.
2. Patients should have stage III or IV disease, staged T3-4 and/or N2-3, M0
3. Patients must have a Karnofsky performance status of >= 70
4. Age >/= 18 years
5. No hematogenous metastatic disease
6. Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC) of > 1500 cells/mm**3 and platelet count of > 100,000 cells/mm**3; adequate hepatic function with total bilirubin <= Upper Limit of Normal (ULN), aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) may be up to 2.5 times the upper limit of normal if alkaline phosphatase is normal. Alkaline phosphatase may be up to 4 * ULN if aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) are normal. Patients who have SGPT > 1.5 ULN and alkaline phosphatase > 2.5 * ULN are not eligible.
7. Creatinine clearance > 50 ml/min determined by 24 hour collection or nomogram: CrCl male = (140 - age) * (weight as kg)/serum Cr * 72 CrCl female = 0.85 * (CrCl male)
8. Patients must not have received previous surgery, other than diagnostic biopsy, or radiation, for this cancer. Patients may have received neoadjuvant chemotherapy which must have been completed > 3 weeks from beginning therapy on this trial.
9. Patients with a history of non-melanoma skin cancer, or other previous malignancies treated 5 years or more prior to the current tumor from which the patient has remained continually disease-free, are eligible.
10. Patients must sign a study-specific informed consent form.
11. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for 6 months thereafter. Childbearing potential will be defined as women who have had menses within the past 12 months, who have not had tubal ligation or bilateral oophorectomy.

Exclusion Criteria:

1. Histology other than squamous cell carcinoma.
2. Evidence of metastases (below the clavicle or distant) by clinical or radiographic means.
3. Karnofsky performance status < 70
4. Prior therapy with inhibitors of epidermal growth factor receptor (EGFR)
5. Prior radiotherapy to the head and neck
6. Patients with simultaneous primaries
7. Patients with a past history of malignancy (excluding non melanoma skin cancers, and cancers treated > 5 years prior for which patient remains continuously disease free).
8. Pregnant/breast-feeding women are ineligible.
9. Patients refusing or unable to sign the informed consent.
10. Patients with pre-existing peripheral neuropathy NCI Common Toxicity Criteria (CTC) grade 2 or worse.
11. Patients with a history of severe hypersensitivity reaction to Taxotere® and/or Polysorbate 80 must be excluded.
12. Patients may not use ketoconazole, St. John's Wort, or erythromycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of erlotinib and docetaxel during concomitant boost radiation | 6 weeks of treatment, followed
  MTD defined as highest dose level in which 6 patients have been treated with less than or equal to 2 instances of Dose-limiting toxicity (DLT) from 2 sources: 1) Out-of-field toxicity from unirradiated sites secondary to systemic therapy(erlotinib and docetaxel); 2) In-field toxicity from irradiated sites secondary to combined treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org